CLINICAL TRIAL: NCT01582451
Title: A Comparison of LY2605541 Versus Insulin Glargine Alone or in Combination With Pre-study Oral Antihyperglycemic Medications in Patients With Type 2 Diabetes Mellitus Previously Treated With Basal Insulin: An Open-Label, Randomized Study The IMAGINE 5 Study
Brief Title: A Study of LY2605541 in Participants With Type 2 Diabetes Mellitus
Acronym: IMAGINE 5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14703; I2R-MC-BIDJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Results first posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LY2605541; basal insulin peglispro; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LY2605541 (Experimental): Administered by subcutaneous (SQ) injection once daily at bedtime. Initial dose based on dose of prestudy basal insulin and adjusted based on fasting blood glucose (FBG). LY2605541 will be given alone or in combination with up to 3 pre-study oral antihyperglycemic medications (OAMs) whose use is not excluded in combination with insulin. Treatment may last up to 52 weeks.
  Interventions: Drug: LY2605541
- Insulin glargine (Active Comparator): Administered by SQ injection once daily at bedtime. Initial dose based on dose of prestudy basal insulin and adjusted based on FBG. Insulin glargine will be used alone or in combination with up to 3 pre-study OAMs whose use is not excluded in combination with insulin. Treatment may last up to 52 weeks.
  Interventions: Drug: Insulin glargine

INTERVENTIONS:
Drug: LY2605541
  Other Names: Insulin peglispro
  Arms: LY2605541
Drug: Insulin glargine
  Arms: Insulin glargine

SUMMARY:
The purpose of this study is to compare LY2605541 and insulin glargine using the following measures after participants have been treated for 26 weeks:

* Change in participants' overall blood sugar control
* The rate of night time low blood sugar episodes
* The number of participants that reach blood sugar targets without low blood sugar episodes at night
* The rate of low blood sugar episodes reported over a 24-hour period

ELIGIBILITY:
Inclusion Criteria:

* Have had type 2 diabetes mellitus for at least 1 year
* Have been receiving basal insulin (neutral protamine Hagedorn [NPH], detemir, or glargine) and a stable dose of 0 to 3 oral antihyperglycemic medications (OAMs) used as specified in the local prescribing information for at least 90 days prior to screening. At least 1 of the OAMs must be dosed at, or above, half the maximum daily dose allowed by local regulations or at the maximally tolerated dose
* Have a hemoglobin A1c (HbA1c) less than or equal to 9.0% at screening
* Have a body mass index (BMI) less than or equal to 45.0 kilograms per square meter (kg/m^2)
* Women of childbearing potential who are not breastfeeding, have a negative pregnancy test at screening and randomization, do not plan to become pregnant during the study, and have practiced reliable birth control for at least 6 weeks prior to screening and will continue to do so during the study and until 2 weeks after the last dose of study drug

Exclusion Criteria:

* Have routinely used insulin glargine twice daily in the 90 days prior to the study or have used routine, mealtime insulin therapy (outside of pregnancy) anytime in the past 6 months, except for short-term treatment up to a maximum of 4 continuous weeks
* Have used rosiglitazone, pramlintide, glucagon-like peptide 1 (GLP-1) receptor agonist concurrently or within 90 days prior to screening
* For participants on OAMs: have any restrictions for cardiac, renal, and hepatic diseases in the local product regulations
* Are taking, or have taken within the 90 days preceding screening, prescription or over-the-counter medications to promote weight loss
* Have had any episodes of severe hypoglycemia within 6 months prior to screening
* Have had 1 or more episodes of diabetic ketoacidosis or hyperosmolar state/coma in the 6 months prior to screening
* Have cardiac disease with functional status that is New York Heart Association Class III or IV
* Have a history of renal transplantation, or are currently receiving renal dialysis or have serum creatinine greater than or equal to 2 milligrams per deciliter (mg/dL) (177 micromoles per liter [µmol/L])
* Have obvious clinical signs or symptoms of liver disease (excluding non-alcoholic fatty liver disease [NAFLD]), acute or chronic hepatitis, non-alcoholic steatohepatitis (NASH), or elevated liver enzyme measurements
* Have had a blood transfusion or severe blood loss within 3 months prior to screening or have known hemoglobinopathy, hemolytic anemia, or sickle cell anemia, or any other traits of hemoglobin abnormalities known to interfere with the measurement of HbA1c
* Have active or untreated cancer, have been in remission from clinically significant cancer(other than basal cell or squamous cell skin cancer) for less than 5 years, or are at increased risk for developing cancer or a recurrence of cancer in the opinion of the investigator
* Are receiving chronic (lasting longer than 14 consecutive days) systemic glucocorticoid therapy (excluding topical, intranasal, intraocular, and inhaled preparations) or have received such therapy within the 8 weeks immediately preceding screening
* Have fasting triglycerides greater than 400 mg/dL (4.5 millimoles per liter [mmol/L]) at screening
* Have an irregular sleep/wake cycle (for example, participants who sleep during the day and work during the night) in the investigator's opinion
* Lipid-lowering medication: Are using or have used any of the following:

  * niacin preparations as a lipid-lowering medication and/or bile acid sequestrants within 90 days prior to screening or
  * lipid-lowering medication at a dose that has not been stable for at least 90 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT -5 hours, EST), Study Director — Eli Lilly and Company
Locations (61):
- United States (33):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mesa, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Port Richey, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oviedo, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roswell, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Crystal Lake, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloomington, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangor, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rockville, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raleigh, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Akron, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Delaware, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jackson, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Round Rock, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bountiful, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Federal Way, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olympia, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milwaukee, Wisconsin
- Czechia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beroun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brandýs nad Labem
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aschaffenburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Mergentheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Damme
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rhaunen
- Greece (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chalcis
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Israel (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Acre
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beersheba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Holon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nazareth
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Raanana
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bayamón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
- Romania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oradea
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sibiu
- Russia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arkhangelsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Novosibirsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alzira
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cadiz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palma de Mallorca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pozuelo de Alarcón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Teruel

REFERENCES:
- [Derived] Qu Y, White RD, Ruberg SJ. Accurate Collection of Reasons for Treatment Discontinuation to Better Define Estimands in Clinical Trials. Ther Innov Regul Sci. 2023 May;57(3):521-528. doi: 10.1007/s43441-022-00491-0. Epub 2022 Dec 21. PMID 36542287
- [Derived] Sanyal A, Cusi K, Hartman ML, Zhang S, Bastyr EJ 3rd, Bue-Valleskey JM, Chang AM, Haupt A, Jacober SJ, Konrad RJ, Zhang Q, Hoogwerf BJ. Cytokeratin-18 and enhanced liver fibrosis scores in type 1 and type 2 diabetes and effects of two different insulins. J Investig Med. 2018 Mar;66(3):661-668. doi: 10.1136/jim-2017-000609. Epub 2017 Nov 21. PMID 29167192
- [Derived] Orchard TJ, Cariou B, Connelly MA, Otvos JD, Zhang S, Antalis CJ, Ivanyi T, Hoogwerf BJ. The effects of basal insulin peglispro vs. insulin glargine on lipoprotein particles by NMR and liver fat content by MRI in patients with diabetes. Cardiovasc Diabetol. 2017 Jun 6;16(1):73. doi: 10.1186/s12933-017-0555-1. PMID 28587667
- [Derived] Cusi K, Sanyal AJ, Zhang S, Hartman ML, Bue-Valleskey JM, Hoogwerf BJ, Haupt A. Non-alcoholic fatty liver disease (NAFLD) prevalence and its metabolic associations in patients with type 1 diabetes and type 2 diabetes. Diabetes Obes Metab. 2017 Nov;19(11):1630-1634. doi: 10.1111/dom.12973. Epub 2017 Jun 22. PMID 28417532
- [Derived] Buse JB, Rodbard HW, Trescoli Serrano C, Luo J, Ivanyi T, Bue-Valleskey J, Hartman ML, Carey MA, Chang AM; IMAGINE 5 Investigators. Randomized Clinical Trial Comparing Basal Insulin Peglispro and Insulin Glargine in Patients With Type 2 Diabetes Previously Treated With Basal Insulin: IMAGINE 5. Diabetes Care. 2016 Jan;39(1):92-100. doi: 10.2337/dc15-1531. Epub 2015 Nov 17. PMID 26577417

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2605541: LY2605541 was administered by subcutaneous (SQ) injection once daily at bedtime for up to 52 weeks. Initial dose based on dose of prestudy basal insulin and adjusted based on fasting blood glucose (FBG).
- Insulin Glargine: Insulin glargine was administered by SQ injection once daily at bedtime for up to 52 weeks. Initial dose based on dose of prestudy basal insulin and adjusted based on FBG.
Period: Overall Study
Arm/Group | LY2605541 | Insulin Glargine
Started | 307 | 159
Received at Least 1 Dose of Study Drug | 305 | 159
Completed | 275 | 139
Not Completed | 32 | 20
Not completed — Adverse Event | 1 | 3
Not completed — Death | 3 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 11 | 3
Not completed — Withdrawal by Subject | 13 | 9
Not completed — Physician Decision | 3 | 0
Not completed — Sponsor Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- LY2605541: LY2605541 was administered by SQ injection once daily at bedtime for up to 52 weeks. Initial dose based on dose of prestudy basal insulin and adjusted based on FBG.
- Total: Total of all reporting groups
Arm/Group | LY2605541 | Insulin Glargine | Total
Number analyzed (Participants) | 307 | 159 | 466
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.84 (8.52) | 60.38 (10.10) | 61.34 (9.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 66 | 198
  Male | 175 | 93 | 268
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 57 | 25 | 82
  Not Hispanic or Latino | 215 | 115 | 330
  Unknown or Not Reported | 35 | 19 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 17 | 9 | 26
  White | 280 | 148 | 428
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 170 | 85 | 255
  Czechia | 20 | 10 | 30
  Greece | 16 | 5 | 21
  Spain | 27 | 12 | 39
  Romania | 16 | 14 | 30
  Israel | 16 | 8 | 24
  Russia | 17 | 9 | 26
  Germany | 25 | 16 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 26-week Endpoint in Hemoglobin A1c (HbA1c)
Description: HbA1c is a test that measures a participant's average blood glucose level over a 2 to 3 month timeframe. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for stratification factors (country, baseline low-density lipoprotein cholesterol [LDL-C, <100 milligrams per deciliter (mg/dL) and ≥100 mg/dL], and sulfonylurea (SU) or meglitinide use), visit, treatment, visit-by-treatment interaction, and baseline HbA1c.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable HbA1c data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 302 | 157
percentage of HbA1c | -0.82 (0.04) | -0.29 (0.06)

2. Secondary Outcome: Change From Baseline to 52 Weeks in HbA1c
Description: LS means were calculated using MMRM adjusting for stratification factors (country, baseline LDL-C [<100 mg/dL and ≥100 mg/dL], and SU or meglitinide use), visit, treatment, visit-by-treatment interaction, and baseline HbA1c.
Time Frame: Baseline, 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 302 | 157
percentage of HbA1c | -0.67 (0.05) | -0.22 (0.06)

3. Secondary Outcome: Rate of Total and Nocturnal Hypoglycemia Events (Adjusted by 30 Days)
Description: Hypoglycemic episodes are defined as events which are associated with reported signs and symptoms of hypoglycemia and/or documented blood glucose (BG) concentrations of ≤70 mg/dL (3.9 millimoles per liter [mmol/L]). A nocturnal hypoglycemic event occurred between bedtime and waking. Group mean rates of total and nocturnal hypoglycemia (per 30 days) are presented and were calculated from negative binomial regression models (number of episodes = treatment + baseline hypoglycemia rate + baseline SU or meglitinide use, with log [exposure in days/30] as an offset variable). Group Mean is estimated by taking the inverse link function on individual participant covariates first and then averages over all participants.
Time Frame: Baseline through 26 weeks and Baseline through 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: events/participant/30 days
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 304 | 159
events/participant/30 days
  Total hypoglycemia, 0-26 weeks | 1.55 (0.13) | 1.98 (0.19)
  Total hypoglycemia, 0-52 weeks | 1.24 (0.10) | 1.62 (0.15)
  Nocturnal hypoglycemia, 0-26 weeks | 0.43 (0.06) | 1.04 (0.15)
  Nocturnal hypoglycemia, 0-52 weeks | 0.35 (0.06) | 0.88 (0.14)

4. Secondary Outcome: Percentage of Participants That Have Total and Nocturnal Hypoglycemic Events
Description: Hypoglycemic episodes are defined as events which are associated with reported signs and symptoms of hypoglycemia and/or documented BG concentrations of ≤70 mg/dL (3.9 mmol/L). A nocturnal hypoglycemic event occurred between bedtime and waking. The percentage of participants was calculated by dividing the number of participants with hypoglycemic episodes by the total number of participants analyzed, multiplied by 100.
Time Frame: Baseline through 26 weeks and Baseline through 52 weeks
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 304 | 159
percentage of participants
  Total hypoglycemia, 0-26 weeks | 76.3 | 80.5
  Total hypoglycemia, 0-52 weeks | 80.3 | 83.0
  Nocturnal hypoglycemia, 0-26 weeks | 46.1 | 62.3
  Nocturnal hypoglycemia, 0-52 weeks | 50.3 | 67.3

5. Secondary Outcome: Percentage of Participants With HbA1c Equal to or Less Than (≤) 6.5% and Less Than (<) 7.0%
Description: The percentage of participants was calculated by dividing the number of participants reaching target HbA1c by the total number of participants analyzed, multiplied by 100.
Time Frame: 26 and 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable HbA1c data. Missing endpoints were imputed with by applying the last observation carried forward (LOCF) method to the post-baseline data.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 302 | 157
percentage of participants
  HbA1c ≤6.5%, 26 weeks | 50.3 | 28.7
  HbA1c ≤6.5%, 52 weeks | 43.4 | 28.0
  HbA1c <7.0%, 26 weeks | 72.5 | 52.2
  HbA1c <7.0%, 52 weeks | 63.9 | 45.9

6. Secondary Outcome: Percentage of Participants With HbA1c <7.0% and Without Nocturnal Hypoglycemia
Description: Hypoglycemic episodes are defined as an event which is associated with reported signs and symptoms of hypoglycemia and/or a documented blood glucose concentration of ≤70 mg/dL (3.9 mmol/L). A nocturnal hypoglycemic event occurred between bedtime and waking. The percentage of participants was calculated by dividing the number of participants with HbA1c <7.0% without nocturnal hypoglycemia by the total number of participants analyzed, multiplied by 100.
Time Frame: 26 and 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable HbA1c data. Missing endpoints were imputed with by applying the LOCF method to the post-baseline data.
Measure: Number; unit: percentage of participants
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 302 | 157
percentage of participants
  26 weeks | 40.1 | 18.5
  52 weeks | 34.8 | 10.2

7. Secondary Outcome: Fasting Serum Glucose (FSG) (by Laboratory)
Description: LS means were calculated using MMRM adjusting for stratification factors (country, baseline HbA1c [≤8.0% and >8.0%], baseline LDL-C [<100 mg/dL and ≥100 mg/dL], and SU or meglitinide use), visit, treatment, visit-by-treatment interaction, and baseline FSG.
Time Frame: 26 and 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable FSG data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 302 | 157
milligrams per deciliter (mg/dL)
  26 weeks | 103.80 (1.88) | 119.50 (2.64)
  52 weeks | 107.61 (1.94) | 115.74 (2.72)

8. Secondary Outcome: Fasting Blood Glucose (FBG) (by Self Monitoring)
Description: LS means were calculated using MMRM adjusting for stratification factors (country, baseline HbA1c [≤8.0% and >8.0%], baseline LDL-C [<100 mg/dL and ≥100 mg/dL], and SU or meglitinide use), visit, treatment, visit-by-treatment interaction, and baseline FBG.
Time Frame: 26 and 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable FBG data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 303 | 158
milligrams per deciliter (mg/dL)
  26 weeks | 106.32 (1.08) | 104.50 (1.51)
  52 weeks | 110.61 (1.19) | 107.46 (1.68)

9. Secondary Outcome: Intra-participant Variability in Fasting Blood Glucose (FBG)
Description: FBG was measured by self-monitored blood glucose (SMBG). Between-day glucose variability is measured by the standard deviation of FBG. LS means were calculated using MMRM adjusting for the stratification factors (country, baseline HbA1c [≤8.5% and >8.5%], baseline LDL-C [<100 mg/dL and ≥100 mg/dL], and SU or meglitinide use), treatment, visit, treatment-by-visit interaction, and baseline FBG intra-participant variability.
Time Frame: 26 and 52 weeks
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 302 | 158
mg/dL
  26 weeks | 13.70 (0.57) | 17.90 (0.80)
  52 weeks | 14.18 (0.65) | 17.38 (0.91)

10. Secondary Outcome: 6-point Self-monitored Blood Glucose (SMBG)
Description: SMBG measurements were taken at 6 time points (pre-morning meal [fasting], pre-midday meal, pre-evening meal, bedtime, approximately 0300 hours, and pre-morning meal [fasting] on the next day) and were performed on 2 non-consecutive days in the week prior to next office visit. LS means were calculated using MMRM adjusting for stratification factors (baseline HbA1c [≤8.5% and >8.5%], country, LDL-C [<100 mg/dL and ≥100 mg/dL], and SU or meglitinide use), visit, treatment, visit-by-treatment interaction, and baseline BG values.
Time Frame: 26 and 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable SMBG data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 288 | 148
mg/dL
  Pre-morning meal, 26 weeks | 107.93 (1.30) | 104.11 (1.83)
  Pre-midday meal, 26 weeks: number analyzed (Participants) | 287 | 145
  Pre-midday meal, 26 weeks | 120.87 (2.20) | 132.56 (3.11)
  Pre-evening meal, 26 weeks: number analyzed (Participants) | 287 | 146
  Pre-evening meal, 26 weeks | 125.87 (2.18) | 141.45 (3.08)
  Bedtime, 26 weeks: number analyzed (Participants) | 285 | 143
  Bedtime, 26 weeks | 146.54 (2.61) | 161.48 (3.69)
  0300 hours, 26 weeks: number analyzed (Participants) | 281 | 142
  0300 hours, 26 weeks | 118.43 (2.04) | 120.42 (2.87)
  Pre-morning meal next day, 26 weeks | 106.28 (1.36) | 102.79 (1.90)
  Pre-morning meal, 52 weeks | 110.84 (1.39) | 108.22 (1.94)
  Pre-midday meal, 52 weeks: number analyzed (Participants) | 287 | 145
  Pre-midday meal, 52 weeks | 121.34 (2.17) | 130.55 (3.06)
  Pre-evening meal, 52 weeks: number analyzed (Participants) | 287 | 146
  Pre-evening meal, 52 weeks | 128.53 (2.00) | 141.31 (2.82)
  Bedtime, 52 weeks: number analyzed (Participants) | 285 | 143
  Bedtime, 52 weeks | 146.92 (2.37) | 161.83 (3.34)
  0300 hours, 52 weeks: number analyzed (Participants) | 281 | 142
  0300 hours, 52 weeks | 122.23 (1.96) | 121.07 (2.76)
  Pre-morning meal next day, 52 weeks | 110.38 (1.41) | 106.68 (1.97)

11. Secondary Outcome: HbA1c
Description: as for outcome 2
Time Frame: 26 and 52 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 302 | 157
percentage of HbA1c
  26 weeks | 6.60 (0.04) | 7.13 (0.06)
  52 weeks | 6.75 (0.05) | 7.20 (0.06)

12. Secondary Outcome: Insulin Dose Per Kilogram of Body Weight
Description: Daily basal insulin dose is presented. LS means were calculated using MMRM adjusting for the stratification factors (country, baseline HbA1c [≤8.5% and >8.5%], baseline LDL-C [<100 mg/dL and ≥100 mg/dL], and SU or meglitinide use), treatment, visit, treatment-by-visit interaction, and baseline insulin dose.
Time Frame: 26 and 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable insulin dose data.
Measure: Least Squares Mean (Standard Error); unit: units per kilogram per day (U/kg/day)
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 304 | 159
units per kilogram per day (U/kg/day)
  26 weeks | 0.57 (0.01) | 0.49 (0.01)
  52 weeks | 0.58 (0.01) | 0.49 (0.02)

13. Secondary Outcome: Number of Insulin Dose Adjustments to Steady-state
Description: The number of dose adjustments required to reach a steady dose is presented. LS means were calculated from negative binomial regression models, where the number of dose adjustments = treatment + stratification factors (country, baseline HbA1c [≤8.5% and >8.5%], baseline LDL-C [<100 mg/dL and ≥100 mg/dL], and SU or meglitinide use).
Time Frame: Baseline through 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable insulin dose data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: number of dose adjustments
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 304 | 159
number of dose adjustments | 4.06 (0.16) | 2.75 (0.20)

14. Secondary Outcome: European Quality of Life - 5 Dimension (EuroQol-5D) Score
Description: The EuroQol-5D is a generic, multidimensional, health-related, quality-of-life instrument. The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a 3-level scale of 1-3 (no problem, some problems, and extreme problems). These combinations of attributes are converted into a weighted health-state Index Score according to the United States population-based algorithm. Scores range from -0.11 to 1.0, where a score of 1.0 indicates perfect health. LS means were calculated using an analysis of covariance (ANCOVA) model adjusting for treatment, stratification factors (country, baseline HbA1c [≤8.5% and >8.5%], and SU or meglitinide use), and baseline EuroQol-5D score.
Time Frame: 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable EuroQol-5D data at both baseline and post-baseline. Missing endpoints were imputed by applying the LOCF method to the post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 290 | 146
units on a scale | 0.87 (0.01) | 0.88 (0.01)

15. Secondary Outcome: Insulin Treatment Satisfaction Questionnaire (ITSQ) Score
Description: ITSQ is a validated instrument containing 22 items that assess treatment satisfaction for participants with diabetes and on insulin. The questionnaire measures satisfaction from the following 5 domains: Inconvenience of Regimen, Lifestyle Flexibility, Glycemic Control, Hypoglycemic Control, Insulin Delivery Device. Data presented are the transformed overall score on a scale of 0-100, where a higher score indicate better treatment satisfaction. LS means were calculated using ANCOVA with treatment and stratification factors (country, baseline HbA1c [≤8.5% and >8.5%], and SU or meglitinide use) as fixed effects and baseline value of the ITSQ score as a covariate.
Time Frame: 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable ITSQ data at both baseline and post-baseline. Missing endpoints were imputed by applying the LOCF method to the post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 291 | 148
units on a scale | 85.69 (0.63) | 84.43 (0.89)

16. Secondary Outcome: Adult Low Blood Sugar Survey (LBSS) Score
Description: LBSS (also referenced as Hypoglycemia Fear Survey - II [HFS-II]) is a 33-item questionnaire that measures 1) behaviors to avoid hypoglycemia and its negative consequences (15 items) and 2) worries about hypoglycemia and its negative consequences (18 items). Responses are made on a 5-point Likert scale where 0 = Never and 4 = Always. Total score is the sum of all items (range 0-132). Higher total scores reflect greater fear of hypoglycemia. LS means were calculated using ANCOVA with treatment and stratification factors (country, baseline HbA1c [≤8.5% and >8.5%], and SU or meglitinide use) as fixed effects and baseline value of the LBSS score as a covariate.
Time Frame: 26 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable LBSS data at both baseline and post-baseline. Missing endpoints were imputed by applying the LOCF method to the post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 292 | 148
units on a scale | 16.57 (0.77) | 15.63 (1.08)

17. Secondary Outcome: Change From Baseline in Body Weight
Description: LS means were calculated using MMRM adjusting for stratification factors (country, baseline HbA1c [≤8.5% and >8.5%], LDL-C [<100 mg/dL and ≥100 mg/dL, except for the LDL-C outcome variable], and SU or meglitinide use), visit, treatment, visit-by-treatment interaction, and baseline body weight.
Time Frame: Baseline, 26 weeks, 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable body weight data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 303 | 157
kilograms (kg)
  26 weeks | 0.50 (0.17) | 0.94 (0.24)
  52 weeks | 0.69 (0.23) | 1.32 (0.32)

18. Secondary Outcome: Change From Baseline in Lipid Profile
Description: Concentrations of cholesterol, high-density lipoprotein cholesterol (HDL-C), LDL-C, and triglycerides are summarized. LS means were calculated using MMRM adjusting for stratification factors (country, baseline HbA1c [≤8.5% and >8.5%], LDL-C [<100 mg/dL and ≥100 mg/dL, except for the LDL-C outcome variable], and SU or meglitinide use), visit, treatment, visit-by-treatment interaction, and baseline value of corresponding lipid outcome variable.
Time Frame: Baseline, 26 weeks, 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable lipid data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 302 | 157
mg/dL
  Cholesterol, 26 weeks | 2.24 (1.60) | 3.70 (2.25)
  Cholesterol, 52 weeks | -1.35 (1.63) | 2.78 (2.29)
  HDL-C, 26 weeks | -1.74 (0.37) | -0.06 (0.52)
  HDL-C, 52 weeks | -3.52 (0.37) | -2.01 (0.51)
  LDL-C, 26 weeks | -0.05 (1.43) | 4.54 (2.00)
  LDL-C, 52 weeks | -3.38 (1.45) | 3.41 (2.03)
  Triglycerides, 26 weeks | 22.53 (3.73) | -2.90 (5.23)
  Triglycerides, 52 week | 27.39 (4.00) | 12.02 (5.59)

19. Secondary Outcome: Number of Participants With Change in Anti-LY2605541 Antibodies
Description: The number of participants with a treatment-emergent anti-LY2605541 antibody response (TEAR) is summarized. TEAR is defined as change from baseline to post-baseline in the anti-LY2605541 antibody level either from undetectable to detectable, or from detectable to the value with at least 130% relative increase from baseline.
Time Frame: Baseline through 52 weeks
Population: Participants who were randomized, had at least 1 dose of study medication, and had evaluable anti-LY2605541 antibody data at baseline and post-baseline.
Measure: Number; unit: participants
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 301 | 157
participants | 70 | 30

ADVERSE EVENTS:
Description: Includes events from participants who were randomized and had at least 1 dose of study medication.
Arm/Group | LY2605541 | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 36/305 | 22/159
Other Adverse Events (participants affected / at risk) | 223/305 | 104/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2605541 (N=305) | Insulin Glargine (N=159)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (5)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (3) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 1 (2) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Cardiac vein perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 2 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/131 (1) | 0/66 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/174 (0) | 1/93 (1)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Urethral obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/174 (2) | 0/93 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/131 (0) | 1/66 (1)
Prostatitis (Reproductive system and breast disorders) | 1/174 (1) | 0/93 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1/131 (1) | 0/66 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (10) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2605541 (N=305) | Insulin Glargine (N=159)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 19 (21) | 6 (6)
Nausea (Gastrointestinal disorders) | 12 (13) | 4 (7)
Bronchitis (Infections and infestations) | 14 (14) | 5 (5)
Influenza (Infections and infestations) | 13 (14) | 11 (13)
Nasopharyngitis (Infections and infestations) | 50 (63) | 27 (33)
Sinusitis (Infections and infestations) | 18 (19) | 9 (9)
Upper respiratory tract infection (Infections and infestations) | 16 (18) | 8 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (18) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 21 (22) | 9 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7) | 9 (9)
Dizziness (Nervous system disorders) | 7 (8) | 5 (6)
Headache (Nervous system disorders) | 15 (21) | 12 (27)
Anxiety (Psychiatric disorders) | 2 (5) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 9 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (8)
Rash (Skin and subcutaneous tissue disorders) | 10 (11) | 1 (1)
Hypertension (Vascular disorders) | 8 (8) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days